CLINICAL TRIAL: NCT00738296
Title: Vytorin on Carotid Intima-media Thickness and Overall Rigidity
Acronym: VYCTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alejandra Meaney Martinez, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Regional 1o de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008_018; MK0653A-164
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin; Pravastatin

ARMS (3):
- A (Active Comparator): Group A: Comparator
  Interventions: Drug: simvastatin
- B (Active Comparator): Group B: Comparator
  Interventions: Drug: pravastatin
- C (Experimental): Group C: Drug
  Interventions: Drug: ezetimibe (+) simvastatin

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Patients will receive the combination of ezetimibe/simvastatin 10/20 mg o.d. with the possibility to increase the dose to 10/40 mg o.d. for 1 year. Tablets
  Other Names: MK0653A; Vytorin
  Arms: C
Drug: simvastatin — Patients will receive 40mg od. With the possibility to escalate the dose to 80 mg o.d. if therapeutic goals not attained; for 1 year. Tablets
  Other Names: Zocor
  Arms: A
Drug: pravastatin — Patients will receive pravastatin 40 mg o.d. with the possibility to add up 10mg of ezetimibe daily if LDL-C goal is not achieved; for 1 year. Tablets
  Arms: B

SUMMARY:
Comparison of the effect on the progression of the carotid intima-media interphase thickness (GIM), arterial rigidity according to the measurement of the pulse wave speed and direct measurement of the carotid and aortic rigidities and an inflammation marker (PCR) in patients with established cardiovascular disease (myocardial infarct, atherosclerotic coronary disease), diabetes mellitus type 2 or equivalent risk of coronary disease and a low density lipoprotein level > 100 mg/dL, treated with simvastatin, pravastatin or the combination of simvastatin-ezetimibe during a period of at least one year.

ELIGIBILITY:
Inclusion Criteria:

* Ldl-C Levels >100 Mg/Dl
* Patients Who Have Signed The Consent
* Patients Of ages between 30 and 75 Years Old
* Patients Of Both Genders
* Patients With Established Cardiovascular Disease, Diabetes With Or Without Established Cardiovascular Disease
* Patients Without Previous Treatment With Ezetimibe

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The annual progression of the slope of the maximum average GIM and the arterial rigidity. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Meaney, MD, PhD, Principal Investigator — Hospital Regional 1o de Octubre, ISSSTE